CLINICAL TRIAL: NCT06145620
Title: Effects of a Prehabilitation Program Based on Therapeutic Exercise, Back Care Education and Neuroscience Pain Education in Patients Undergoing Lumbar Radiculopathy Surgery
Brief Title: Effects of a Prehabilitation Program in Patients Undergoing Lumbar Radiculopathy Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, ARGUISUELAS MARTINEZ MARÍA DOLORES, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEEI23/459
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic exercise, back care and pain neuroscience education group (Experimental)
  Interventions: Other: Physiotherapy
- Standarized written exercise group (Active Comparator)
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — The intervention involves the visualization of different videos explaining the performance of lumbar strengthening exercises, measures for back care, and neuroscience pain education.

SUMMARY:
The purpose of the following study is to analyze the effects of a prehabilitation program based on therapeutic exercise, back care education and pain neuroscience education through the visualization of videos, compared to standardized written therapeutic exercise in patients undergoing lumbar radiculopathy surgery.

DETAILED DESCRIPTION:
So far, there are no previous studies that analyze the effects of a prehabilitation program including therapeutic exercise, back care education and pain neuroscience education through the visualization of videos in patients undergoing lumbar radiculopathy surgery.

This is a multicenter randomized clinical trial aimed at analyzing the effects of a 4 weeks prehabilitation program based on video visualization versus the performance of standardized written exercises in patients undergoing lumbar radiculopathy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older, diagnosed with lumbar radiculopathy, and scheduled for surgery. The symptoms will be predominantly leg pain with or without neurological deficit, with surgical decompression justified.

Exclusion Criteria:

* Patients currently receiving any other non-pharmacological treatment or physical therapy for the management of lumbar radiculopathy.
* Proposed for surgery with instrumentation (e.g., spinal fusion, arthrodesis).
* Suffering from a chronic pain-related condition (e.g., fibromyalgia, chronic fatigue syndrome).
* Symptoms of spinal cord compression.
* Diagnosed with a malignant tumor.
* Mental illness.
* Previously undergone spinal surgery.
* No access to any internet-enabled device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 4 weeks
  Disability score (0-100). Higher score indicates higher disability.

SECONDARY OUTCOMES:
SF-McGill Pain Questionnaire (SF-MGPQ) | 4 weeks
  Pain score (0-45). Higher score indicates higher pain level
Numerical Rating Scale (NRS) | 4 weeks
  Pain score 0-10. Higher score indicates higher pain intensity.
EuroQol-5D (EQ-5D) | 4 weeks
  Quality of life score (-0.5 to 1).Higher score indicates higher health-related quality of life
Fear avoidance beliefs questionnaire (FABQ) | 4 weeks
  FABQ-Work subscale (ranging from 0 to 42) and FABQ-Physical Activity subscale (ranging from 0 to 24). Higher score indicates more signs of fear avoidance
Hospital Anxiety and Depression Scale (HADS) | 4 weeks
  Anxiety and depression score (0-21). Hhigher score indicates greater symptoms of anxiety and depression.
Pain catastrophizing scale (PCS) | 4 weeks
  pain catastrophizing score (0-52). Higher scores indicate greater pain catastrophizing
Tampa scale for kinesiophobia (TSK-11SV) | 4 weeks
  kinesiophobia score (11-44). Higher scores indicate greater kinesiophobia
International Physical Activity Questionnaire (IPAQ) | 4 weeks
  Physical activity level (MET minutes a week). Higher scores indicate higher physical activity level

CONTACTS AND LOCATIONS:
Locations (1):
- Arguisuelas Martinez Maria Dolores, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindback Y, Tropp H, Enthoven P, Abbott A, Oberg B. PREPARE: presurgery physiotherapy for patients with degenerative lumbar spine disorder: a randomized controlled trial. Spine J. 2018 Aug;18(8):1347-1355. doi: 10.1016/j.spinee.2017.12.009. Epub 2017 Dec 15. PMID 29253630
- [Background] Louw A, Butler DS, Diener I, Puentedura EJ. Development of a preoperative neuroscience educational program for patients with lumbar radiculopathy. Am J Phys Med Rehabil. 2013 May;92(5):446-52. doi: 10.1097/PHM.0b013e3182876aa4. PMID 23478459
- [Background] Goudman L, Huysmans E, Ickmans K, Nijs J, Moens M, Putman K, Buyl R, Louw A, Logghe T, Coppieters I. A Modern Pain Neuroscience Approach in Patients Undergoing Surgery for Lumbar Radiculopathy: A Clinical Perspective. Phys Ther. 2019 Jul 1;99(7):933-945. doi: 10.1093/ptj/pzz053. PMID 30921465